CLINICAL TRIAL: NCT06071923
Title: Effect of Thyroid Disorders in Metabolic Fatty Liver Changes
Brief Title: Effect of Thyroid Disorders in Liver Diseases
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Tasneem Mohammed Ali, Principal investigator, Assiut University
Other Study IDs: 04-2023-200396
Record Dates: First submitted 2023-10-02; First posted 2023-10-10 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Fibroscan — Scan the liver for metabolic fatty changes

SUMMARY:
Aims of the Research

1. To detect correlation between hyperthyroidism and non alcoholic fatty liver disease (NAFLD).
2. To detect hepatic risk in subclinical and clinical hypothyroidism .
3. To detect early liver disorders in thyroid disorders using fibroscan .

DETAILED DESCRIPTION:
Non alcoholic fatty liver disease (NAFLD) has been a health problem of growing significance all over the world; its prevalence is increasing in both developed and developing countries ,the overall prevalence of NAFLD worldwide was estimated to be 32.4%.prevalence increased significantly over time.

considering the increasing incidence of NALAD/NASH, especially in developed and developing countries, it is anticipated that cirrhosis due to these conditions may exceed other causes of cirrhosis in a near future..

Thyroid gland is involved in energy homeostasis, lipid and carbohydrate metabolism, regulation of body weight and adipogenesis.

In a clinical setting, subclinical hypothyroidism has been associated with metabolic syndrome, cardiovascular mortality and disturbance of lipid metabolism.

The prevalence of hypothyroidism was reported to 16.8% among patients with NAFLD/NASH.

In recent years, growing body of evidence has led to speculation on the association between NAFLD/NASH and thyroid dysfunction.

Therefore, understanding the pathophysiology, risk factors and new treatment options of NAFLD/NASH should be among the priorities in the field of hepatology

ELIGIBILITY:
Inclusion Criteria:

* The study will include thyroid patients over one year duration ( age above 18 years old

Exclusion Criteria:

1. History of liver failure or patient known to have congenital liver disease.
2. Medications associated with weight gain .
3. Patients who have diabetes mellitus.
4. patients who already have liver disease eg; chronic viral hepatitis, liver cirrhosis.
5. Patients on antistatin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with thyroid disorders and age above 18 years
Sampling Method: Non-Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Detect correlation between hyperthyroid diseases and NASH . | Baseline
  Test the patients of thyroid disorders for metabolic fatty liver changes